CLINICAL TRIAL: NCT01004419
Title: Phase I Trial of Vandetanib (ZD6474, Zactima) and Fulvestrant (Faslodex) as Third-Line Treatment of Advanced Non-Small Cell Lung Cancer
Brief Title: Trial of ZD6474 and Faslodex in Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Support for investigational products has been withdrawn.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: AstraZeneca (Industry); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2008-0009; CO 07505
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: non small cell lung cancer; vandetanib; ZD6474; fulvestrant; faslodex; phase 1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib plus fulvestrant (Experimental): vandetanib by mouth once daily for 28 days plus fulvestrant intra-muscular injection each cycle
  Interventions: Drug: ZD6474 (vandetanib); Drug: Faslodex (Fulvestrant)

INTERVENTIONS:
Drug: ZD6474 (vandetanib) — vandetanib (100 mg or 200 mg or 300 mg) by mouth once daily for 28 days
  Other Names: ZD6474, Zactima
Drug: Faslodex (Fulvestrant) — Fulvestrant 500 mg intra-muscular injection on Day 1 and 250 mg Day 15 of cycle 1 Cycles 2 and beyond: Fulvestrant 500 mg intra-muscular injection on Day 1, every 28 days.
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of vandetanib and fulvestrant; to find the maximum tolerated dose of these two drugs; and to evaluate response rate and assess toxicity of this combination.

DETAILED DESCRIPTION:
Current treatment for metastatic non-small cell lung cancer (NSCLC) is inadequate, with a median survival of 8-12 months. Second-line therapy options include cytotoxic agents or molecularly-targeted agents such as erlotinib. Nevertheless, only 7-9% of patients will respond to standard second-line treatment. Treatment-related side effects from cytotoxic drugs and declining performance status in patients with progressing disease are significant issues in this patient population. Novel approaches with molecularly-targeted agents are clearly needed.

The combination of vandetanib and fulvestrant addresses the potential to interfere with multiple interdependent growth-stimulatory pathways simultaneously. Recent work has revealed cross-talk between epidermal growth factor receptor (EGFR) and estrogen receptor (ER) pathways. This clinical trial will evaluate the clinical interaction of the EGFR inhibitor, vandetanib, in combination with the ER down-regulator, fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically/histologically confirmed non-small cell lung cancer (NSCLC), advanced (stage IIIB w/ effusion or IV).
* Performance status of 0, 1, or 2
* Brain metastases must be clinically stable after treatment with surgery and/or radiotherapy
* Must have received two prior systemic anti-cancer regimens for recurrent/ metastatic disease, including one platinum-containing regimen
* Prior radiotherapy, chemotherapy and/or treatment with investigational agents is allowed provided that the patient has recovered from the treatment-related side effects to grade ≤1, and that at least 3 weeks has passed since the last dose
* Required laboratory values demonstrating adequate bone marrow, kidney, liver, and blood clotting function.
* Negative pregnancy test for women of childbearing potential within 7 days prior to study entry
* Life expectancy of 3 months or more
* Must tolerate intramuscular injections
* No prior or concurrent use of estrogen replacement therapy
* No concurrent use of cytotoxic, immunologic, hormonal, or investigational agent intended for the antitumor treatment of NSCLC

Exclusion Criteria:

* Prior therapy with any anti-EGFR therapy such as gefitinib (IRESSA), erlotinib (TARCEVA), vandetanib (ZD6474, ZACTIMA), or fulvestrant (FASLODEX), or an aromatase inhibitor
* Clinically significant cardiac event such as myocardial infarction, superior vena cava syndrome, New York Heart Association (NYHA) classification of heart disease ≥ 2 within 3 months before entry
* History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation), which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia
* Presence of left bundle branch block
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age
* History of QTc prolongation as a result from other medications that required discontinuation of that medication
* QTc with Bazett's correction that is unmeasurable, or ≥ 480 msec on screening ECG
* Potassium <4.0 mmol/L despite supplementation, or potassium above the CTCAE grade 1 upper limit
* Serum calcium above the CTCAE grade 1 upper limit
* Magnesium below the normal range despite supplementation, or above the CTCAE grade 1 upper limit
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
* Diagnosis of active interstitial lung disease
* Currently active diarrhea that may affect drug absorption
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and basal cell or squamous cell carcinoma of the skin
* Concomitant use of medications that are potent inducers of CYP3A4 are not allowed within 2 weeks of study or during the study
* Any unresolved toxicity greater than CTC grade 1 from previous anti-cancer therapy
* Major surgery within 4 weeks, or incompletely healed surgical incision
* Women who are currently pregnant or breast feeding
* History of bleeding diathesis (ie, disseminated intravascular coagulation [DIC], clotting factor deficiency)
* History of hypersensitivity to active or inactive excipients of fulvestrant (ie castor oil or Mannitol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Toleration of combination of fulvestrant/vandetanib | Monthly

SECONDARY OUTCOMES:
Response rate to combination of fulvestrant/vandetanib | End of trial
Safety of combination of fulvestrant/vandetanib | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Tien Hoang, M.D., Principal Investigator — University of Wisconsin, Madison